CLINICAL TRIAL: NCT04824768
Title: Immediate Effects of Tecar Therapy on Spasticity and Functionality of the Lower Limb in Chronic Post-stroke Survivors.
Brief Title: Effect of Tecar in Addition of Functional Massage in Post-stroke Spasticity
Acronym: Tecar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Rosa Cabanas Valdés, PhD, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRet 1
Record Dates: First submitted 2021-03-27; First posted 2021-04-01 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Stroke Sequelae; Massage; Spasticity, Muscle; Electrotherapy
Keywords: Stroke; Spasticity; Tecar therapy; Functional massage; Muscle tone; Capacitive Resistive Electric Transfer Therapy (CRet)
MeSH Terms: conditions — Muscle Spasticity; Stroke

STUDY DESIGN:
Intervention Model Description: An introductory massage was performed on the lumbar region and hamstrings of the most affected leg, in conjunction with Tecar therapy in the resistive modality (80W). Functional Massage was then performed on the gastrocnemius, with Tecar in resistive mode (100-120W), and then in capacitive mode (180-200VA).
Who Masked: Participant, Outcomes Assessor
Masking Description: An introductory massage was performed on the lumbar region and hamstrings of the most affected leg, in conjunction with Tecar therapy in the resistive modality (0W). Functional Massage was then performed on the gastrocnemius, with Tecar in resistive mode (0W), and then in capacitive mode (0VA).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 30 min session of Tecar Therapy with functional massage on the rectus femoris, and gastrocnemius. Tecar therapy in the resistive modality (80W) on lower back and hamstrings and in rectus femoris and gastrocnemius with resistive mode (100-120W), and then in capacitive mode(180-200VA)
  Interventions: Device: Tecar Therapy
- Control group (Sham Comparator): 30 min session of Tecar Therapy with functional massage on the rectus femoris, and gastrocnemius. Sham stimulation was provided by only turn on the device but dose is 0.
  Interventions: Device: Sham Tecar Therapy

INTERVENTIONS:
Device: Tecar Therapy — CRet is a non-invasive diathermy technique that provides high frequency energy generating a thermal effect on soft tissues. Functional massage (FM) is a non-invasive manual therapy technique that combines rhythmical passive joint mobilization with compression of the muscular belly with the muscle-tendon insertions to be treated.
  In prone position, subjects will get a 7 min preparation massage with CRet on resistive mode (80-100W), on the lumbar area, followed by a 5 min preparation massage with CRet on resistive mode (100-120 W) on the hamstrings. Then a 5 min F.M with passive ankle dorsiflexion and CRet on resistive mode (110-120 W) will be performed on the gastrocnemius medialis and lateralis, followed by a 4 min FM with CRet on capacitive mode (180-250VA) on the mentioned area.
  In supine position, a 5 min FM with passive knee flexion and CRet on resistive mode 8.
  A physiotherapist will monitor the temperature of the patient's treated area every 2 minutes
  Arms: Experimental group
Device: Sham Tecar Therapy — In prone position, subjects will get a 7 min preparation massage with CRet on resistive mode (0 W), on the lumbar area, followed by a 5 min preparation massage with CRet on resistive mode (0 W) on the hamstrings. Then a 5 min FM with passive ankle dorsiflexion and CRet on resistive mode (0 W) will be performed on the gastrocnemius medialis and lateralis, followed by a 4 min FM with CRet on capacitive mode (0 VA) on the mentioned area.
  In supine position, a 5 min FM with passive knee flexion and CRet on resistive mode 0.
  A physiotherapist will monitor the temperature of the patient's treated area every 2 minutes
  Arms: Control group

SUMMARY:
Spasticity is due to an abnormal processing of a normal input from muscle spindles in the spinal cord.

DETAILED DESCRIPTION:
Stroke often affects sensory-motor networks and descending tracts, as reflected by several signs of upper motor neuron syndrome. One symptom is post-stroke spasticity. It is due to an abnormal processing of a normal input from muscle spindles in the spinal cord. It is often defined by a velocity-dependent increase in muscle tone and a resistance to passive muscle stretch. It has neural (increased reflex activity) and non-neural (altered visco-elastic properties due to immobilization) components. The prevalence of spasticity ranges from 25%-43% at 6 months post-stroke. Chronic spasticity can decrease the number of sarcomeres. As a result, the proportion of connective tissue in the muscle and fasciae can increase. These subjects present fibrosis that have augmented passive muscle stiffness due to structural and functional adaptations inside the muscle cells. Soft tissue changes may cause the pulling forces to be transmitted more readily to the muscle spindles, which can intensify sensory input thus increasing spasticity. It has a potential impact on lower limb function, which affects passive muscle stretch, range of motion, and motor unit recruitment during voluntary contraction. In the stance phase of gait, the deformity also produces an inadequate base of support, which is associated with balance impairments. This increases the risk of falls, reduces patient participation in daily activities, and decreases health-related quality of life. Physiotherapy treatments of spasticity aim to decrease excessive muscular tone, ease mobility, give the patient the sense of right position and avoid joint limitations.

Functional massage is a non-invasive manual therapy technique that combines rhythmical passive joint mobilization with compression and decompression of the muscular belly with the tendinomuscular insertions to treat. It is indicated in cases of muscle stiffness associated with pain.

Tecar therapy or Capacitive Resistive Electric Transfer Therapy (CRet) is a non-invasive diathermy technique which provides high frequency energy (300 KHz-1.2 MHz) generating a thermal effect on soft tissues. CRet is used to facilitate tissue regeneration, and it does not need a surface-cooling system, as its wave frequency is lower than in conservative diathermy. CRet effectiveness has been evaluated in several studies. It is effective in the treatment of chronic musculoskeletal disorders, where a temperature increase on deep tissues is needed in order to generate changes on its viscoelasticity. This effect may be beneficial in the spasticity treatment since spasticity onset and development may be affected by structural changes in muscular and tendinous fibers.

No studies on the effects of CRet in post-stroke spasticity treatment were found.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Stroke
* Scoring 1 on the Modified Ashworth Scale (MAS) for hip or/and knee flexion or/and ankle dorsiflexion on the most affected limb
* Scoring 25 or plus on the Montreal Cognitive Assessment (MoCA)

Exclusion Criteria:

* Having suffered a traumatism on the lower limbs three months, or less, before the intervention
* Suffer other neurological disease
* Presence of osteosynthetic material
* Pacemaker wearing
* Treatment with botulinum toxin or another antispastic medication, six months , or less, before the intervention
* Carry baclofen pump
* Functional inability to adopt the prone or supine position on the treatment table
* Functional inability to sit, stand and walk
* Poor language and communication skills that make difficult to understand the informed consent
* Contraindications to Functional Massage (infectious diseases, inflammatory vascular conditions, acute inflammation, hemorrhagic, fever)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Muscle tone | T1: Baseline, T2: Immediately after treatment and T3: follow up 30 minutes after treatment
  To evaluate the immediate changes in terms of muscle tone on the rectus femoris, medialis and gastrocnemius after one session with CRet as coadjuvant of functional massage by modified Ashworth Scale of Hip flexion-extension, knee flexion-extension, ankle plantar flexion and dorsiflexion. The minimum and maximum values are 0 and 4, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Muscle stiffness | T1: Baseline, T2: Immediately after treatment and T3: follow up 30 minutes after treatment
  To evaluate muscle stiffness on rectus femoris and gastrocnemius after one session with CRet as coadjuvant of functional massage by mioton Myoton Pro, Myoton Ltds., Estonia) on the muscular belly.
Muscle flexibility | T1: Baseline, T2: Immediately after treatment and T3: follow up 30 minutes after treatment
  Myoton-Pro device applied on the muscle belly of rectus femoris, internal and external gastrocnemius
Muscle relaxation | T1: Baseline, T2: Immediately after treatment and T3: follow up 30 minutes after treatment
  Myoton-Pro device applied on the muscle belly of rectus femoris, internal and external gastrocnemius
Passive range of motion | T1: Baseline, T2: Immediately after treatment and T3: follow up 30 minutes after treatment
  Goniometry applied on passive hip flexion and extension, passive knee flexion and ankle plantar flexion and dorsiflexion with a wedge under the knees. The force applied by the physiotherapist will be recorded with a goniometer and will be applied to the head of the metatarsals.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa C Cabanas-Valdés, PhD, Principal Investigator — Universitat Internacional de Catalunya
Locations (2):
- Spain (2):
  - Universitat Internacional de Catalunya, Barcelona, Catalonia
  - Laura Garcia Rueda, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Francisco GE, McGuire JR. Poststroke spasticity management. Stroke. 2012 Nov;43(11):3132-6. doi: 10.1161/STROKEAHA.111.639831. Epub 2012 Sep 13. No abstract available. PMID 22984012
- [Background] Gillard PJ, Sucharew H, Kleindorfer D, Belagaje S, Varon S, Alwell K, Moomaw CJ, Woo D, Khatri P, Flaherty ML, Adeoye O, Ferioli S, Kissela B. The negative impact of spasticity on the health-related quality of life of stroke survivors: a longitudinal cohort study. Health Qual Life Outcomes. 2015 Sep 29;13:159. doi: 10.1186/s12955-015-0340-3. PMID 26415945
- [Background] Lopez-de-Celis C, Hidalgo-Garcia C, Perez-Bellmunt A, Fanlo-Mazas P, Gonzalez-Rueda V, Tricas-Moreno JM, Ortiz S, Rodriguez-Sanz J. Thermal and non-thermal effects off capacitive-resistive electric transfer application on the Achilles tendon and musculotendinous junction of the gastrocnemius muscle: a cadaveric study. BMC Musculoskelet Disord. 2020 Jan 20;21(1):46. doi: 10.1186/s12891-020-3072-4. PMID 31959172
- [Background] Clijsen R, Leoni D, Schneebeli A, Cescon C, Soldini E, Li L, Barbero M. Does the Application of Tecar Therapy Affect Temperature and Perfusion of Skin and Muscle Microcirculation? A Pilot Feasibility Study on Healthy Subjects. J Altern Complement Med. 2020 Feb;26(2):147-153. doi: 10.1089/acm.2019.0165. Epub 2019 Oct 3. PMID 31580698
- [Background] Beltrame R, Ronconi G, Ferrara PE, Salgovic L, Vercelli S, Solaro C, Ferriero G. Capacitive and resistive electric transfer therapy in rehabilitation: a systematic review. Int J Rehabil Res. 2020 Dec;43(4):291-298. doi: 10.1097/MRR.0000000000000435. PMID 32909988
- [Result] Rehme AK, Grefkes C. Cerebral network disorders after stroke: evidence from imaging-based connectivity analyses of active and resting brain states in humans. J Physiol. 2013 Jan 1;591(1):17-31. doi: 10.1113/jphysiol.2012.243469. Epub 2012 Oct 22. PMID 23090951
- [Result] Trompetto C, Marinelli L, Mori L, Pelosin E, Curra A, Molfetta L, Abbruzzese G. Pathophysiology of spasticity: implications for neurorehabilitation. Biomed Res Int. 2014;2014:354906. doi: 10.1155/2014/354906. Epub 2014 Oct 30. PMID 25530960
- [Result] Zorowitz RD, Gillard PJ, Brainin M. Poststroke spasticity: sequelae and burden on stroke survivors and caregivers. Neurology. 2013 Jan 15;80(3 Suppl 2):S45-52. doi: 10.1212/WNL.0b013e3182764c86. PMID 23319485
- [Result] Lance JW. The control of muscle tone, reflexes, and movement: Robert Wartenberg Lecture. Neurology. 1980 Dec;30(12):1303-13. doi: 10.1212/wnl.30.12.1303. No abstract available. PMID 7192811
- [Result] Stecco C, Porzionato A, Lancerotto L, Stecco A, Macchi V, Day JA, De Caro R. Histological study of the deep fasciae of the limbs. J Bodyw Mov Ther. 2008 Jul;12(3):225-30. doi: 10.1016/j.jbmt.2008.04.041. Epub 2008 Jun 13. PMID 19083678
- [Result] Lieber RL, Runesson E, Einarsson F, Friden J. Inferior mechanical properties of spastic muscle bundles due to hypertrophic but compromised extracellular matrix material. Muscle Nerve. 2003 Oct;28(4):464-71. doi: 10.1002/mus.10446. PMID 14506719
- [Result] Kuo C, Hu G. Post-stroke spasticity: A review of epidemiology, pathophysiology, and treatments. International Journal of Gerontology. 2018;12(4):280-284.
- [Result] Cacho RdO, Cacho EWA, Loureiro AB, et al. The spasticity in the motor and functional disability in adults with post-stroke hemiparetic. Fisioterapia em Movimento. 2017;30(4):745-752.